CLINICAL TRIAL: NCT03246555
Title: A Randomized, Double-blind, Active-controlled, 2-parallel Group, Optional Titration, Multicenter, Phase 3b Study to Evaluate the Efficacy and Safety of Fimasartan Versus Perindopril Monotherapy With and Without Diuretics Combination in Elderly Patients With Essential Hypertension
Brief Title: Fimasartan in the Senior Subjects
Acronym: FITNESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR-FMS-CT-304
Record Dates: First submitted 2017-07-25; First posted 2017-08-11 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: The Elderly (≥ 70 Years) With Essential Hypertension
MeSH Terms: interventions — fimasartan; Hydrochlorothiazide; Perindopril; Indapamide

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fimasartan or Fimasartan/Hydrochlorothiazide (Experimental)
  Interventions: Drug: Fimasartan or Fimasartan/Hydrochlorothiazide
- Perindopril or Perindopril/Indapamide (Active Comparator)
  Interventions: Drug: Perindopril or Perindopril/Indapamide

INTERVENTIONS:
Drug: Fimasartan or Fimasartan/Hydrochlorothiazide — The treatment in this clinical study starts with fimasartan 30 mg; if blood pressure is not controlled (siSBP ≥ 140 mmHg or siDBP ≥ 90 mmHg), the dose is escalated once gradually, and then a diuretic combination is administered. The escalation of dose and administration of diuretic combination are decided after checking blood pressure 4 weeks after the administration of each investigational product.
  Arms: Fimasartan or Fimasartan/Hydrochlorothiazide
Drug: Perindopril or Perindopril/Indapamide — The treatment in this clinical study starts with penrindopril 2.5 mg; if blood pressure is not controlled (siSBP ≥ 140 mmHg or siDBP ≥ 90 mmHg), the dose is escalated once gradually, and then a diuretic combination is administered. The escalation of dose and administration of diuretic combination are decided after checking blood pressure 4 weeks after the administration of each investigational product.
  Arms: Perindopril or Perindopril/Indapamide

SUMMARY:
The objective of this study is to confirm the noninferiority of the blood pressure lowering effect of fimasartan and evaluate its safety compared to perindopril in the elderly with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provided a written consent to participate in this clinical study after receiving an explanation of this study
2. Elderly aged 70 years or older
3. At the screening visit (Visit 1), Blood pressure: Mean blood pressure measured 3 times on the selected arm is as below.

   * For treatment-naïve patients who have not taken drugs for hypertension within the last 3 months from the screening visit: Mean siSBP ≥ 140mmHg
   * For patients with essential hypertension who are taking drugs for hypertension: Mean siSBP ≥ 130mmHg
4. At the baseline visit (Visit 2), Blood pressure: Patients with mild to moderate essential hypertension whose mean siSBP measured 3 times on the selected arm is ≥140 mmHg Patients with treatment compliance of ≥70% during the placebo run-in period
5. Capable of understanding written instructions, cooperative, able to participate until the end of the clinical study

Exclusion Criteria:

1. Severe hypertension patients with mean siSBP ≥ 180 mmHg or siDBP ≥ 110 mmHg (office BP) at the screening visit (Visit 1) and the baseline visit (Visit 2) (However, at screening, it is based on the blood pressures measured from both arms, and the patient is excluded if the result from any of the arms falls within the criteria.)
2. Patients with siSBP ≥ 20 mmHg and siDBP ≥ 10 mmHg in the difference between blood pressures in the selected arm at the screening visit (Visit 1)
3. Patients with a history of secondary hypertension and any history suspected of secondary hypertension (but not limited to the following: coarctation of the aorta, primary hyperaldosteronism, renal artery stenosis, Cushing's syndrome, pheochromocytoma, polycystic kidney disease, etc.)
4. Orthostatic hypotension with symptoms
5. Patients with insulin-dependent diabetes mellitus or uncontrolled diabetes mellitus (HbA1c > 9.0% at the screening visit (Visit 1))
6. Patients with a history of malignant tumor, including leukemia and lymphoma, within the past 5 years (however, participation is allowed if it has not recurred for at least 5 years after a tumor surgery)
7. Patients with any chronic inflammatory disease requiring chronic anti-inflammatory treatment, consumption disease, autoimmune disease like rheumatoid arthritis and systemic lupus erythematosus, etc., or connective tissue disease at present or in the past
8. Patients with a history of hypersensitivity reaction to any component of the investigational product and its similar compound Renin-angiotensin system inhibitors, ACE inhibitors, thiazide diuretics and sulfonamides, Yellow 5 (Sunset Yellow FCF), etc.
9. Patients with hyperlipidemia undergoing LDL (low density lipoprotein) apheresis (patients undergoing LDL hemapheresis using a dextran sulfate cellulose)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 241 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Change in siSBP | 8 weeks
  Change in siSBP from baseline after the administration of the investigational product for 8 weeks

SECONDARY OUTCOMES:
Change in siSBP | Weeks 4, 16 and 24
  Change in siSBP from baseline at Weeks 4, 16 and 24
Change in siDBP | Weeks 4, 8, 16 and 24
  Change in siDBP from baseline at Weeks 4, 8, 16 and 24
Blood pressure response rate | 4, 8 and 16 weeks
  Blood pressure response rate (siSBP < 140 mmHg, or decrease of △siSBP ≥ 20 mmHg after the administration for 4, 8 and 16 weeks compared to baseline) and blood pressure normalization rate after the administration of the investigational products for 4, 8 and 16 weeks(siSBP<140mmHg and siDBP<90mmHg)
Change from baseline in the differences in standing SBP and DBP compared to their sitting measurements | 4, 8, 16 and 24 weeks
  Change from baseline in the differences in standing SBP and DBP compared to their sitting measurements after the administration of the investigational product for 4, 8, 16 and 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang, Seoul, South Korea

REFERENCES:
- [Derived] Lee HY, Kim KI, Ihm SH, Rhee MY, Sohn IS, Park S, Jeon ES, Song JM, Pyun WB, Sung KC, Kim MH, Kim SH, Kim SY, Kim SJ, Kim EJ, Shin J, Lee SY, Chun KJ, Jeong JO, Chae SC, Yoo KD, Choi YJ, Park YH, Kim CH. A Randomized, Double-blind, Active-controlled, Two Parallel-Group, Optional Titration, Multicenter, Phase IIIb Study to Evaluate the Efficacy and Safety of Fimasartan Versus Perindopril Monotherapy With and Without a Diuretic Combination in Elderly Patients With Essential Hypertension. Clin Ther. 2021 Oct;43(10):1746-1756. doi: 10.1016/j.clinthera.2021.08.003. Epub 2021 Sep 7. PMID 34503866
- [Derived] Kang MG, Kim KI, Ihm SH, Rhee MY, Sohn IS, Lee HY, Park S, Jeon ES, Song JM, Pyun WB, Sung KC, Kim MH, Kim SH, Kim SY, Kim SJ, Kim EJ, Shin J, Lee SY, Chun KJ, Jeong JO, Chae SC, Yoo KD, Choi YJ, Park YH, Kim CH. Fimasartan versus perindopril with and without diuretics in the treatment of elderly patients with essential hypertension (Fimasartan in the Senior Subjects (FITNESS)): study protocol for a randomized controlled trial. Trials. 2019 Jul 1;20(1):389. doi: 10.1186/s13063-019-3466-5. PMID 31262348